CLINICAL TRIAL: NCT04465032
Title: The Effect of Consecutive Fecal Microbiota Transplantation on Non-Alcoholic Fatty Liver Disease (NAFLD) - a Randomized-controlled Trial -
Brief Title: The Effect of Consecutive Fecal Microbiota Transplantation on Non-Alcoholic Fatty Liver Disease (NAFLD)
Acronym: NAFTx
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Donor Feces Bank (Unknown); Vedanta Biosciences (Unknown)
Responsible Party: Principal Investigator, metushuizen, Principle investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE17-05
Record Dates: First submitted 2020-01-08; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial, randomization 1:1 to allogenic and autologous gut microbiome transplantation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded RCT, randomization by Dutch Donor Feces Bank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous gut microbiome transplantation (Active Comparator): Three autologous (own) fecal transplantations (at baseline, 3 and 6 weeks)
  Interventions: Other: Gut microbiome transplantation
- Allogenic gut microbiome transplantation (Experimental): Three allogenic (lean donor) fecal transplantations (at baseline, 3 and 6 weeks)
  Interventions: Other: Gut microbiome transplantation

INTERVENTIONS:
Other: Gut microbiome transplantation — Fecal transplantation will be performed at baseline and at week 3 and 6. At the Department of Clinical Bacteriology either the autologous or allogenic feces is prepared for donation by an experienced lab co-worker. The fecal transplantation will be performed via gastroduodenal endoscopy at the Department of Gastroenterology by an experienced endoscopist. To alleviate the procedure, midazolam is offered to the participants. Following placement of the endoscope in the horizontal duodenum, 150 mL feces solution is inserted via the endoscope.
  Other Names: Fecal transplantation

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a disease of alarmingly increasing prevalence, linked to metabolic, cardiovascular and malignant morbidity and without any officially approved treatment. It is increasingly recognized that the gut microbiome is implicated in the pathogenesis and progression of numerous chronic diseases, including NAFLD. Through the so-called gut-liver axis, the liver is exposed to gut-bacterial-derived products, including toxins (lipopolysaccharides), enzymes (methylamines), alcohol, and short-chain fatty acids (mainly acetate, propionate, and butyrate), that may lead to accumulation of triglycerides, inflammatory responses, oxidative stress and accompanying damage to the hepatocytes. The primary objective is to study the effect of consecutive FMT on liver fat accumulation measured by Magnetic Resonance Images (MRI) LiverMultiscan at 12 weeks. Secondary objectives are weight, waist, blood pressure, metabolic parameters (including glucose, cholesterol, pancreatic beta-cell function, HOMA-IR), objective and subjective stress indicators, gut-microbiota and bile composition and liver enzymes. Stool samples will be collected for microbiota analysis at time point 0, 3, 6 and 12 weeks.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a disease of alarmingly increasing prevalence, linked to metabolic, cardiovascular and malignant morbidity and without any officially approved treatment. It is increasingly recognized that the gut microbiome is implicated in the pathogenesis and progression of numerous chronic diseases, including NAFLD. Through the so-called gut-liver axis, the liver is exposed to gut-bacterial-derived products, including toxins (lipopolysaccharides), enzymes (methylamines), alcohol, and short-chain fatty acids (mainly acetate, propionate, and butyrate), that may lead to accumulation of triglycerides, inflammatory responses, oxidative stress and accompanying damage to the hepatocytes. The investigators hypothesize that altered gut microbiota underlie (hepatic) insulin resistance and liver fat accumulation in NAFLD patients. Fecal microbiota transplantation, through amelioration of gut-microbiota released products like lipopolysaccharides, short-chain fatty acids, alcohol and enzymes, and changes in bile acids, may positively affect NAFLD.

During the study 20 patients will be randomized for infusion of allogenic (lean donor) or autologous (own) feces by gastroscopy at time points 0, 3 and 6 weeks on a 1:1 basis. Prior to randomization, and at 12 weeks, all patients will undergo LiverMultiscan to non-invasively quantify liver fat accumulation and other features of NAFLD. In addition, various metabolic parameters (lipids, HOMA-IR), objective and subjective stress indicators, gut-microbiota and bile composition, and liver enzymes will be measured.

The primary objective is to study the effect on consecutive FMT on liver fat accumulation measured by Magnetic Resonance Images (MRI) LiverMultiscan at 12 weeks. Secondary objectives are alterations in anthropometrical data (weight, waist, blood pressure), changes in fecal microbiota, liver enzymes, bile composition and metabolic parameters including glucose, lipids, pancreatic beta-cell function and insulin resistance measured as HOMA-IR and objective and subjective stress indicators.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI > 27 kg/m2)
* Males and postmenopausal females
* Aged 18 to 70 years
* Hepatic steatosis defined as increased hyperechogenicity of the liver on abdominal ultrasound and/or histological signs of steatosis
* Written informed consent

Exclusion Criteria:

* Exclusion criteria for MRI (claustrophobia, pacemaker, metal implants, etc)
* Any other liver disease than NAFLD/NASH
* Present excessive alcohol use defined as > 2 units/day
* Recent use (< 3 months) of antibiotics
* use of possible drugs interfering microbiota or recent (< 3 months) changes in dosages
* use of GLP-1 RA or SU-derivatives
* Recent (< 3 months) weight change (>5%)
* Cardiovascular co-morbidity defined as heart failure, coronary insufficiency and hypertension in past history
* Previous use of glucocorticosteroids, hormonal substitution, pagitaxel, theofyllin, amiodarone, myelosuppresive agents.
* A psychiatric, addictive or any other disorder that compromises the subjects ability to understand the study content and to give written informed consent for participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the effect on consecutive FMT on liver fat accumulation | 12 weeks
  measured by MRI Livermultiscan

SECONDARY OUTCOMES:
alterations in anthropometric data | 3, 6 and 12 weeks
  differences in weight in kilograms
alterations in anthropometric data | 3, 6 and 12 weeks
  differences in systolic and diastolic blood pressure in mmHg
alterations in anthropometric data | 3, 6 and 12 weeks
  differences in waist in centimeters
alterations in pancreatic beta-cell function and insulin resistance | 3, 6 and 12 weeks
  measured by plasma C-peptide in nmol/L derived during OGTT + arginin
alterations in pancreatic beta-cell function and insulin resistance | 3, 6 and 12 weeks
  measured by glucose in mmol/L derived during OGTT + arginin
alterations in pancreatic beta-cell function and insulin resistance | 3, 6 and 12 weeks
  measured by insulin in mU/L derived during OGTT + arginin
alterations in liver enzymes | 3, 6 and 12 weeks
  Aspartaat aminotransferase (ASAT), alanine aminotransferase (ALAT), gamma glutamyl transpeptidase (GGT), alkalic phosphatase (AF), bilirubin
change in bile composition | 3 and 6 weeks
  measured using endoscopic bile samples (qualitative measurements)
change in bacterial species in small intestine and feces | 3 and 6 weeks
  measured by endoscopic duodenal biopsies and fecal samples
changes in lipid homeostasis | 3, 6 and 12 weeks
  cholesterol, HDL, LDL, triglycerides
alterations in psychological stress | 0 and 12 weeks
  by measuring cortisol levels in hair samples
alterations in psychological stress | week 1, week 4, week 7, week 9 during 7 days
  by reporting psychological stress daily using stress diaries on a scale from 1-10 (non-validated scale)
alterations in psychological stress | 0 and 12 weeks
  by Perceived Stres Scale (PSS) questionnaires, scores on a scale from 0-40
changes in physical activity | during 14 weeks
  measuring physical activity by steps with FitBit activity tracker
changes in physical activity | during 14 weeks
  measuring physical activity by active minutes with FitBit activity tracker
changes in physical activity | during 14 weeks
  measuring physical activity by heart rate with FitBit activity tracker

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groenewegen B, Ruissen MM, Crossette E, Menon R, Prince AL, Norman JM, Ballieux BEPB, Lamb HJ, Terveer EM, Keller JJ, Tushuizen ME. Consecutive fecal microbiota transplantation for metabolic dysfunction-associated steatotic liver disease: a randomized controlled trial. Gut Microbes. 2025 Dec;17(1):2541035. doi: 10.1080/19490976.2025.2541035. Epub 2025 Aug 4. PMID 40755230